CLINICAL TRIAL: NCT03641885
Title: A Randomized Trial of a Social Media Intervention on Promoting Oral Heath Among Iranian Adolescents
Brief Title: A Social Media Intervention on Promoting Oral Heath Among Iranian Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qazvin University Of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir H Pakpour, Director of Social Determinants of Health Research Center, Qazvin University of Medical Sciences, Qazvin University Of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IR.QUMS.REC.1396.601
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Health Behavior; Adolescent Behavior; Parent-Child Relations
MeSH Terms: conditions — Health Behavior; Adolescent Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mother and adolescents (Experimental): an intervention group in which mothers and adolescents receive the intervention and questionnaires via Telegram social media
  Interventions: Behavioral: mothers and adolescents
- adolescents (Experimental): an intervention group in which adolescents receive the intervention and questionnaires via Telegram social media
  Interventions: Behavioral: adolescents
- active control (Active Comparator): mothers and adolescents are in active control group and only receive the questionnaires
  Interventions: Behavioral: active control

INTERVENTIONS:
Behavioral: mothers and adolescents — The intervention package will be sent to mothers and adolescents via Telegram social media. It contains behavior change techniques targeting outcome expectancy, self-efficacy, action planning, coping planning, and self-monitoring. There will be 3 assessment points in time, baselines, 1 month and six months after interventions.
  Arms: mother and adolescents
Behavioral: adolescents — The intervention package will be sent to only adolescents via Telegram social media. It contains behavior change techniques targeting outcome expectancy, self-efficacy, action planning, coping planning, and self-monitoring. There will be 3 assessment points in time, baselines, 1 month and six months after interventions.
  Arms: adolescents
Behavioral: active control — The active control group receives an information sheet regarding recommendations on oral health behavior via telegram. There will be 3 assessment points in time, with 1 month and six months in between.
  Arms: active control

SUMMARY:
Online social networking sites, such as Telegram, possess a number of useful features that could enhance oral health promotion interventions, including the ability of users to share personal information, which is aggregated and displayed to other users .This study is a longitudinal controlled trial that is designed to investigate the effectiveness of a multi-component intervention on improving oral health in adolescents and their mothers. Participants will be allocated in three groups with a) an intervention group in which mothers and children receive the intervention and questionnaires via Telegram, b) only the children receive the intervention via Telegram and mothers and children receive the questionnaires, and c) mothers and children are in active control group and only receive the questionnaires. The intervention package contains behavior change techniques targeting outcome expectancy, self-efficacy, action planning, coping planning, and self-monitoring. The active control group receives an information sheet regarding recommendations on Oral health behaviors. There will be 3 assessment points in time, baseline, 1 month and 6 months after the interventions.

The primary outcome of this study is to estimate the dyadic mechanisms between mothers and their children regarding improving oral health. Secondary outcome is to investigate whether oral health behavior did improve in the intervention groups in general and also to find the psychological mechanism behind the changes during the time of the study.

ELIGIBILITY:
Inclusion Criteria:

* aged 12 to 16
* possess a smartphone
* able or willing to give informed consent

Exclusion Criteria:

* They are not engaged in other oral-health education or research program.
* They have no physical and/or mental disabilities that will impede their ability to perform their own oral hygiene activities.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 791 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
changes in dental busing behavior using a self-reported questionnaire | baseline, 1 Months, 6 months follow-up
  using a self-reported questionnaire

SECONDARY OUTCOMES:
changes in self efficacy using a self-reported questionnaire | baseline, 1 Months, 6 months follow-up
  self efficacy will be assessed using a self-reported questionnaire with four items. All items are rated on a 5-point scale ranging from 1 (strongly disagree) to 5 (strongly agree)
changes in outcome expectancy | baseline, 1 Months, 6 months follow-up
  outcome expectancy will be assessed using a self-reported questionnaire with three items. All items are rated on a 5-point scale ranging from 1 (strongly disagree) to 5 (strongly agree)
changes in coping planning | baseline, 1 Months, 6 months follow-up
  coping planning will be assessed using a self-reported questionnaire with five items. All items are rated on a 5-point scale ranging from 1 (not true) to 5 (totally true)
changes in action planning | baseline, 1 Months, 6 months follow-up
  action planning will be assessed using a self-reported questionnaire with five items. All items are rated on a 5-point scale ranging from 1 (not true) to 5 (totally true)
changes in risk perception | baseline, 1 Months, 6 months follow-up
  risk perception will be assessed using a self-reported questionnaire with three items. All items are rated on a 5-point scale ranging from 1 (very unlikely) to 5 (very likely)
changes in self-monitoring | baseline, 1 Months, 6 months follow-up
  self-monitoring will be assessed using a self-reported questionnaire with four items. All items are rated on a 5-point scale ranging from 1 (not at all true) to 5 (totally true)
changes in intention | baseline, 1 Months, 6 months follow-up
  Behavioral intention will be assessed using a self-reported questionnaire with four items. All items are rated on a 5-point scale ranging from 1 (strongly disagree) to 5 (strongly agree)
changes in perceived social support | baseline, 1 Months, 6 months follow-up
  perceived social support will be assessed using a self-reported questionnaire with three items. All items are rated on a 5-point scale ranging from 1 (strongly disagree) to 5 (strongly agree)
Changes in Community Periodontal Index (CPI) | baseline, 1 Months, 6 months follow-up
  The CPI scores are rated (0 = healthy gingiva, 1 = gingival bleeding, 2 = calculus, 3 = pocket from 4 to 5 mm, and 4 = pocket ≥6 mm
Changes in Turesky Modification of the Quigley-Hein Plaque Index | baseline, 1 Months, 6 months follow-up
  The amount of plaque on each enamel block for each lingual and buccal surface is rated on a six point Likert-type scale ranging from 0 (no plaque) to 5 (plaque covering two-thirds or more of the crown of the tooth).
Changes in Oral health related quality of life | baseline, 1 Months, 6 months follow-up
  The Pediatric Quality of Life Inventory TM (PedsQLTM) Oral Health Scale is used to examine Oral health related quality of life. The scale comprises five items. All responses are reverse scored and transformed into a 0-100-point scale with higher scores representing better Oral health related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Social Determinants of Health Research Center, Qazvin, Iran